CLINICAL TRIAL: NCT01640236
Title: Flare Measurements in Human Radiation Therapy Patients
Status: Completed | Type: Observational
Sponsor: ChromoLogic, LLC (Industry)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: OCDOS_PRO_110314_02
Record Dates: First submitted 2012-07-10; First posted 2012-07-13 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: The Impact of Whole Body Irradiation on Ocular Flare
Keywords: Ocular flare

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a longitudinal Feasibility Study of a novel non-invasive device in assessing radiation dose exposure in humans. All patients receiving whole body irradiation therapy and meeting all other inclusion/exclusion criteria will receive ocular flare meter measurements and slit-lamp examinations on up to eleven occasions starting prior to the first fractional dose of irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be scheduled to receive whole body irradiation in a dose range from 1.5 to 12Gy.
* Subjects must not have received ocular surgery for at least three months prior to study enrolment.
* Subjects must not have a history of uveitis.
* Subjects must have at least one eye free of cataracts
* Subject age must be greater than 18 years
* Subjects must have the ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Inability to give informed consent
* Cataracts in both eyes
* Subject has received ocular surgery within the prior three months
* Subject has a history of uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients meeting the inclusion/exclusion criteria and receiving whole body irradiation at the UCLA Radiation Oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Ocular flare in radiotherapy patients | Daily measurements for the duration of radiotherapy treatment (expected up to four days from start of treatment)
  Determine if ocular flare meter spectra and/or a slit-lamp eye exam can assess radiation dose exposure in individual human radiotherapy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Michell Kamrava, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Radiation Oncology, Los Angeles, California, United States